CLINICAL TRIAL: NCT02881515
Title: Adverse Neurogenic Actions of Dietary Salt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, William Farquhar, Professor, University of Delaware
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 819183
Record Dates: First submitted 2016-08-15; First posted 2016-08-29 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Diet, Sodium-Restricted

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blood Pressure Reactivity (Experimental): Blood Pressure Responses to a cold pressor test and acute exercise will be assessed. This will be performed while subjects are on a low sodium diet (1000 mg/daily), medium sodium diet (2300 mg/daily), and high sodium diet (7000 mg/daily).
  Interventions: Other: Low Sodium Diet; Other: Medium Sodium Diet; Other: High Sodium Diet
- Blood Pressure Variability (Experimental): Twenty four hour blood pressure variability will be assessed. This will be performed while subjects are on a low sodium diet (1000 mg/daily), medium sodium diet (2300 mg/daily), and high sodium diet (7000 mg/daily).
  Interventions: Other: Low Sodium Diet; Other: Medium Sodium Diet; Other: High Sodium Diet

INTERVENTIONS:
Other: Low Sodium Diet — Ten days of low sodium diet
Other: Medium Sodium Diet — Ten days of a medium sodium diet
Other: High Sodium Diet — Ten days of a high sodium diet

SUMMARY:
Excess dietary salt increases the risk for cardiovascular events, even in people that are not hypertensive. There is some evidence that excess dietary salt exaggerates blood pressure and sympathetic nervous system responses to various perturbations and increases blood pressure variability. This proposal will examine the effects of low, medium, and high salt diets on cardiovascular reactivity and blood pressure variability.

DETAILED DESCRIPTION:
Excess dietary salt causes target organ damage and increases the risk for adverse cardiovascular (CV) events independent of blood pressure (BP). Recent data in salt-resistant, normotensive rodents suggest that high dietary salt enhances the excitability or gain of sympathetic circuits, exaggerates sympathetic and CV responses to various stimuli, and increases BP variability (BPV). There are limited data regarding the impact of dietary salt intake on sympathetic nerve activity (SNA) and CV function in salt-resistant humans as well as the underlying mechanisms contributing to these adverse effects. The long-term goal is to determine how dietary salt adversely affects BP regulation and CV health. The objective of this proposal is to comprehensively evaluate the impact of dietary salt intake on SNA and CV reactivity and BPV in normotensive humans. The investigators have 2 specific aims: 1) Aim 1 will test the hypothesis that high dietary salt increases SNA and CV reactivity in normotensive adults, 2) Aim 2 will test the hypothesis that high dietary salt increases BPV in normotensive adults. The expected outcome is to demonstrate that dietary salt loading increases CV reactivity and BPV through a sympathetic nervous system mechanism that originates in the brain. The proposed research is significant, as these studies will provide empirical evidence that dietary salt intake impacts neurohumoral control of the circulation in salt-resistant humans. The proposed research is innovative because it will identify a novel neurogenic action of dietary salt in human CV regulation.

ELIGIBILITY:
Inclusion Criteria:

* normal blood pressure
* men, Women, minorities
* ECG within normal limits
* screening blood panel within normal limits

Exclusion Criteria:

* high blood pressure (>140/90 mmHg)
* history of cardiovascular disease
* history of cancer
* history of diabetes
* history of kidney disease
* obesity (BMI > 30 kg/m2)
* smoking or tobacco use
* current pregnancy
* nursing mothers
* communication barriers

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Blood Pressure Variability | Day 10 of diet (i.e., after 10 days of low, medium, and high sodium diets; crossover design)
  Standard deviation of systolic blood pressure over 24 hours (mmHg)
Blood Pressure Reactivity - Handgrip exercise | Day 10 of diet (i.e., after 10 days of low, medium, and high sodium diets; crossover design)
  Change in Blood pressure during handgrip exercise (mmHg)

SECONDARY OUTCOMES:
Blood Pressure Reactivity - Cold Pressor test | Day 10 of diet (i.e., after 10 days of low, medium, and high sodium diets; crossover design)
  Change in Blood pressure during a cold pressor test (mmHg)
Sympathetic Responses - Handgrip exercise | Day 10 of diet (i.e., after 10 days of low, medium, and high sodium diets; crossover design)
  Sympathetic outflow (bursts per minute)
Sympathetic Responses - Cold Pressor test | Day 10 of diet (i.e., after 10 days of low, medium, and high sodium diets; crossover design)
  Sympathetic outflow (bursts per minute)

CONTACTS AND LOCATIONS:
Overall Officials: William B Farquhar, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Migdal KU, Babcock MC, Robinson AT, Watso JC, Wenner MM, Stocker SD, Farquhar WB. The Impact of High Dietary Sodium Consumption on Blood Pressure Variability in Healthy, Young Adults. Am J Hypertens. 2020 Apr 29;33(5):422-429. doi: 10.1093/ajh/hpaa014. PMID 32006422